CLINICAL TRIAL: NCT00638547
Title: Intrathecal Enzyme Replacement Therapy For Patients With Mucopolysaccharidosis Type I (Hurler Syndrome)
Brief Title: Intrathecal Enzyme Replacement for Hurler Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT2007-10; 0707M11762 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-03-11; First posted 2008-03-19 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Hurler Syndrome
Keywords: Hurler Syndrome; mucopolysaccharidosis type I; Iduronidase deficiency
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — Iduronidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intent-to-Treat (Experimental): All patients who have received at least one dose of Laronidase.
  Interventions: Drug: IRT Laronidase

INTERVENTIONS:
Drug: IRT Laronidase — Laronidase belongs to a class of drugs called enzyme replacement therapies or ERT that provides people with sufficient quantities of an important enzyme that they cannot create on their own. The main ingredient in laronidase is a protein that is identical to a naturally occurring form of the human enzyme alpha-L-iduronidase. Laronidase replaces the missing enzyme alpha-L-iduronidase and restores sufficient enzyme activity to break down GAG buildup.
  Subjects will receive an infusion of Laronidase into his/her spinal fluid approximately 12 weeks before, 2 weeks before, 100 days after and 6 months after transplant. This procedure is done by lumbar puncture
  Other Names: Aldurazyme

SUMMARY:
This protocol will examine whether the enzyme alpha-L-iduronidase (Laronidase), delivered into the spinal fluid of patients with Hurler syndrome at intervals before and after bone marrow transplant, is a safe and effective approach to slow the neurologic degeneration seen in Hurler patients undergoing transplantation.

DETAILED DESCRIPTION:
Subjects will receive an infusion of Laronidase into his/her spinal fluid approximately 12 weeks before, 2 weeks before, 100 days after and 6 months after transplant. This procedure is done by lumbar puncture (also called a "spinal tap").

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of MPS IH (Hurler syndrome) are candidates for this protocol if they are being considered for hematopoietic stem cell transplantation according the University of Minnesota guidelines.

Exclusion Criteria:

* Patients are less than 6 months old, or older than 3 years of age.
* There is a history of clinically-severe hypersensitivity to Laronidase.
* There is a contraindication for repeated lumbar puncture.
* The family is not willing to undergo the necessary procedures and evaluations inherent in the study.
* Consent has not been signed for participation in the 2004-09 study of intravenous Laronidase administration.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2008-01-02 (Actual); Primary Completion 2017-02-18 (Actual); Study Completion 2018-11-18 (Actual)

PRIMARY OUTCOMES:
To demonstrate the efficacy of intrathecally delivering alpha-L-iduronidase in patients with mucopolysaccharidosis type I in decreasing neurodevelopmental deterioration | 1 year

SECONDARY OUTCOMES:
To determine the safety and toxicity of intrathecally delivering alpha-L-iduronidase in patients with mucopolysaccharidosis type I | 1 year
To determine brain changes with magnetic resonance imaging | 1 and 2 years
To determine neurocognitive changes present in patients with Hurler syndrome | 6, 12, and 24 months
To determine cerebral spinal fluid levels of glycosaminoglycans, cytokines and antibodies to Laronidase at baseline and at each point CSF is obtained | through 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — University of Minnesota Medical Center
Locations (1):
- University of Minnesota, Fairview, Minneapolis, Minnesota, United States